CLINICAL TRIAL: NCT06230315
Title: Direct Visual Examination of Airway Via Flexible Fiberoptic Scope After Cervical Spine Surgery
Brief Title: Visual Examination of Airway Via Flexible Fiberoptic Scope After Cervical Spine Surgery
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 905477-11
Record Dates: First submitted 2018-09-05; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Airway Edema
Keywords: leak test; cervical spine surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cervical spine surgery patients: Patients undergoing multilevel cervical spine surgery at Upstate University hospital

SUMMARY:
Airway swelling and edema after cervical spine surgery(CSS) especially in prone position is the direct cause that prohibits patient from extubation. Anterior cervical discectomy and fusion causes severe peri-vertebral soft tissue swelling that was associated with increased postoperative airway complications.

Facial, lip and tongue edema in combination with the cuff leak test and risk factors are currently served as the bases on whether patient can be extubated after spine surgery. Direct visualization of the larynx and inside trachea post-operatively to assess the airway directly using flexible fiberoptic scope as well as to quantify the degree of airway edema has not been investigated.

Investigators are comparing airway before and after cervical spine surgery for any degree of narrowing in the airway using flexible fiberoptic scope. Investigators are also studying the risk factors affecting the degree of narrowing in the airway if any

DETAILED DESCRIPTION:
Because direct visualization of the airway is the most reliable way for the diagnosing and assessing the degree of laryngeal and trachea edema or swelling, investigators sought to do a study to evaluate the degree of airway edema in adult patients undergoing for CSS using direct visualization via flexible fiberoptic and compare the results pre and post- operatively.

The primary outcome will be severity of larynx and trachea edema after cervical spine surgery.

Secondary outcome will be assessment of reliability of airway leak technique and association between face swelling and airway edema.

18 years old and above, 63 number of patient will be enrolled in the study. Patient enrolled who are under going elective cervical spine surgery.Patients involved in the study will be taken to the OR, after induction and prior to intubation asleep flexible fiberoptic scope will be inserted nasally and video record will be taken above and below the glottis, surgery will be continued as planned.

The primary analysis is to test the association of the severity of the laryngeal and tracheal edema with surgical time and number of levels involved in surgery. Investigators will also perform an exploratory analysis to examine the impact of other potential risk factor, including age, fluids and blood products transfusions, ASA( American Society of Anesthesiology) physical status, facial swelling and cuff leak After conclusion of surgery, and when patients are ready for extubation. Quantitative cuff leak will be done, flexible fiber optic scope will be placed through the endotracheal tube, and at the same time of extubation fiber optic scope will be pulled slowly with the endotracheal tube while recording video until we reach a point that approximate same point video was taken prior to intubation, patients who will remain intubated nasal scope will be placed and video will be taken above the glottis with the endotracheal tube in place, another video will be taken for the airway from inside the endotracheal tube.

Study will be aborted if significant resistance during placement of the fiberoptic scope, nasal bleeding happens or hypoxemia requiring ventilation.

Pictures will be saved on USB device and will be assigned a random code that is non-leading to which videos were taken before surgery and which were taken after surgery. Recording prior to intubation will be done as we are withdrawing the scope out, so the motion will be similar to the motion in the video recorded with extubation, hoping that this will be less leading to the blinded ENT surgeon to which was taken before and which after. Patient that will be kept intubated are not blinded.

Pictures will be then shown to ENT surgeon to assess and compare preoperative and postoperative outcome.

Severity of the laryngeal tracheal edema is classified into mild, moderate, and severe. According to the reduction of the cross-section of the trachea lumen, Mild edema is defined as reduction <30%, Moderate < 50%, severe >50% (8).

ENT surgeon will grade the degree of narrowing in the trachea to:

1. No edema to < 30%
2. 31%-50%
3. > 50%.

And above the trachea into

1. none.
2. mild.
3. severe.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient age 18-70 years.
2. Elective cervical spine surgeries involving in upper CSS, ≥ 2 levels, surgical duration ≥ 2 hours
3. ASA class <4

Exclusion Criteria:

1. RSI (rapid-sequence induction) and patients with high aspiration risk (postpartum).
2. Emergency surgery
3. Angioedema
4. History of airway malignancy.
5. Recent upper airway surgery.
6. Significant recent upper airway infection or abscess.
7. History of radiation therapy
8. Nasogastric tube in place.
9. Tracheostomy in place.
10. History of basal skull fracture or extensive maxillofacial fracture.
11. Severe nasal septum deviation.
12. Morbid obesity BMI > 40.
13. Surgery involves in C1.
14. History of epistaxis or bleeding disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing multilevel cervical spine surgery are recruited as study subjects.
  Inclusion and exclusion criteria as described above
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Degree of airway swelling - subglottic and supraglottic | 24 hours
  Surgical time and number of levels involved in surgery as factors affecting degree of airway swelling.

SECONDARY OUTCOMES:
Degree of airway swelling - subglottic and supraglottic | 24 hours
  Examine the impact of other potential risk factors including age, fluids and blood products transfusions, ASA status, facial swelling and cuff leak.

CONTACTS AND LOCATIONS:
Overall Officials: Luay Nubani, MBCHB, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- Suny Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No